CLINICAL TRIAL: NCT07122349
Title: An Interventional Study to Facilitate the Development of a Cannabis Impairment Detection Device in Adult Cannabis Users
Brief Title: Cannabis Impairment Detection Device Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaize (Industry)
Collaborators: Dicentra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 22-GPHCV-01
Record Dates: First submitted 2025-08-06; First posted 2025-08-14 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Cannabis Intoxication
Keywords: Cannabis; Marijuana; Intoxication; Impairment; Eye Test; Ocular; Drug
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gaize Device (Experimental)
  Interventions: Device: Cannabis Impairment Test

INTERVENTIONS:
Device: Cannabis Impairment Test — Automated Drug Recognition Expert Ocular Tests administered via VR Headset, includes test for Lack of Smooth Pursuit, Horizontal and Vertical Gaze Nystagmus, Lack of Convergence, and Pupillary Rebound Dilation. Tests are preceded by an automated system calibration process.

SUMMARY:
The goal of this study is to develop a cannabis impairment detection device in adult cannabis users. The main question[s] it aims to answer are:

* Is the investigational device accurate and reliable at detecting cannabis impairment?
* is the device safe for the collection of eye movement data from cannabis intoxicated individuals? Participants will be administered a series of Drug Recognition Expert Ocular Tests via the Gaize headset following cannabis consumption.

ELIGIBILITY:
Inclusion Criteria:

* Adults 19, years or older, having given written informed consent to participate in the research trial and certifying that they will not drive for a period of at least 6 hours post discharge.
* Having used cannabis at least one time prior
* Having access to legal cannabis
* Normal or corrected to normal vision using either glasses or contact lenses, or surgery.

Exclusion Criteria:

* Enrolled in, or participated in another clinical trial within 30 days before the study
* Having a prosthetic eye
* Blood pressure greater than 160/90 mmHg and heart rate greater than 100 bpm.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Incidence of device/procedure related Adverse Events/Serious Adverse Events during study intervention | Immediately after testing.
  Number of participants experiencing complications related to the investigational device (headache, dizziness, nausea, etc.)

SECONDARY OUTCOMES:
Drug Recognition Expert Protocol Eye Test Scores | up to 90 minutes
  Correlation between scores at baseline and post cannabis consumption (10 min, 30 min, 60 min, 90 min)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Fichtler, Study Chair — Gaize
Locations (1):
- Dicentra, Toronto, Ontario, Canada